CLINICAL TRIAL: NCT00001996
Title: A Phase II Open Randomized Comparison of 566C80 and Pentamidine Isethionate for the Treatment of Pneumocystis Carinii Pneumonia in AIDS Patients Who Are Intolerant of Trimethoprim / Sulfamethoxazole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 053B; 05
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-05

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Pentamidine; Acquired Immunodeficiency Syndrome; atovaquone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atovaquone; Pentamidine

INTERVENTIONS:
Drug: Atovaquone
Drug: Pentamidine isethionate

SUMMARY:
To compare the safety of atovaquone (566C80) with intravenous (IV) pentamidine for the treatment of mild to moderate Pneumocystis carinii pneumonia (PCP) in AIDS patients who are intolerant of therapy with trimethoprim / sulfamethoxazole (TMP / SMX) by comparing the incidence of premature discontinuation of therapy due to toxicity. To compare the efficacy of 566C80 with intravenous (IV) pentamidine for the treatment of mild to moderate PCP in the same population.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* History of, or are currently experiencing, intolerance to TMP / SMX, or to another sulfonamide, which required discontinuation of therapy.
* Pneumocystis carinii pneumonia (PCP).
* Willing and able to give informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded.

* Malabsorption disorder or vomiting that would, in the judgement of the investigator, potentially limit the retention and absorption of an oral therapy.
* Concurrent bacterial, fungal, or viral pneumonitis, pulmonary Kaposi's sarcoma, or other concurrent illness, or chronic pulmonary disease that, in the investigator's opinion, would make interpretation of drug efficacy difficult.
* Present occurrences of abnormal prolongation of QT interval on standard, 12 lead EKG.

Concurrent Medication:

Excluded:

* Drugs with potential anti-pneumocystis effect (eg:
* sulfonamides, dapsone, trimethoprim, other dihydrofolate reductase (DHFR) inhibitors, primaquine, clindamycin, sulfonylureas).
* Ganciclovir.
* Zidovudine.
* Investigational agents including anti-retroviral agents (ddI, ddC, etc.). Patients receiving these drugs prior to entry must discontinue their use during the therapy phase (21 days) of the trial.
* Corticosteroids (except replacement therapy) during the 21 day treatment period (Strata A and C Patients).
* Class 1A antiarrhythmics (ie:
* quinidine, procainamide, disopyramide).

Patients with the following are excluded:

* Judged by the investigator to be in impending respiratory failure.
* Known intolerance to parenteral pentamidine isethionate, or therapeutic failure with same for treatment of current episode of PCP.
* Significant psychosis or emotional disorder that, in the investigator's opinion, would preclude the patient from adhering to the protocol.
* Inability or unwillingness to take medication orally or with food.
* Prior documented glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* History, or present occurrences, of abnormal prolongation of QT interval on standard, 12 lead EKG.
* Termination from FDA 053A due to toxicity.
* For patients entering under historic intolerance criteria (Groups A and B), prior therapy for this episode of PCP is an exclusion.

Prior Medication:

Excluded:

* Treatment within 4 weeks of entry for a prior episode of PCP.
* For patients entering under historic intolerance criteria (Groups A and B), prior therapy for this episode of PCP is an exclusion.

Required:

* Adjuvant prednisone for patient enrolled in Strata B or D.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - East Bay AIDS Ctr, Berkeley, California
  - Kaiser Foundation Hosp, Harbor City, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - AIDS Community Research Consortium, Redwood City, California
  - Davies Med Ctr, San Francisco, California
  - Dr Patrick Joseph, San Ramone, California
  - Infectious Disease Research Consortium of Georgia, Atlanta, Georgia
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Boston City Hosp, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Gathe, Joseph, M.D., Houston, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Dohn M, Weinberg W, Rosenstock J, Follansbee S, Torres R, Caldwell P. Atovaquone vs. pentamidine for pneumocystis carinii pneumonia in patients with AIDS. Int Conf AIDS. 1993 Jun 6-11;9(1):372 (abstract no PO-B10-1421)